CLINICAL TRIAL: NCT04744324
Title: Effects of Self-supporting Care Model on Activities of Daily Living for Patients With Stroke
Brief Title: Self-supporting Care Model in Home Environment for Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, En-Chi Chiu, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SKH-20201006R
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Activities of Daily Living
Keywords: Stroke; Self-supporting Care Model; Home Care Services
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-supporting Care Group (Experimental): Self-supporting Care in home
  Interventions: Behavioral: Self-supporting Care
- Control group (Active Comparator): Home Health Education
  Interventions: Behavioral: Home health education

INTERVENTIONS:
Behavioral: Self-supporting Care — Individualized self-supporting care with four principals (i.e., drinking water, exercise, excretion, and nutrition)
  Arms: Self-supporting Care Group
Behavioral: Home health education — Individualized home health education
  Arms: Control group

SUMMARY:
The purpose of this study was to administer intervention based on self-supporting care model in home environment and to explore the effects of this intervention on stroke patients' activities of daily living, movement, cognition, nutritional status, and quality of life.

DETAILED DESCRIPTION:
Subjects were randomized to intervention group and control group. The experiment was designed as randomized cross-over control trial. The primary outcome included 8 measures: Barthel Index-based Supplementary Scales, Canadian Occupational Performance Measure, Fugl-Meyer Assessment, Balance Computerized Adaptive Testing, Mini Mental State Examination-2nd edition, Mini Nutritional Assessment, Stroke Impact Scale, and Stroke Self-Efficacy Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* age > 20 years
* Diagnosis of stroke
* The modified Rankin Scale : 2~4
* Keep sitting for half an hour by himself/herself
* Follow instructions
* Willing to sign the subject's consent

Exclusion Criteria:

* Diagnosis of dementia
* History of orthopedic diseases or peripheral nerve injury
* readmission because of stroke

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Barthel Index -based Supplementary Scales | Baseline to 4 weeks
  The Barthel Index-based Supplementary Scales assesses basic activities of daily living using three scales:actual performance, ability, and self-perceived difficulty. The score ranges the three scales (i.e., actual performance, ability, and self-perceived difficulty)is 0-20, 0-18, and 0-20, respectively. A higher score indicates better basic activities of daily living.
Canadian Occupational Performance Measure | Baseline to 4 weeks
  The Canadian Occupational Performance Measure is to measure occupational performance though three areas: self-care, productivity, and leisure. Patients define important activities and classify them with a score of one to 10. A higher score indicates better occupational performance.
Fugl-Meyer Assessment | Baseline to 4 weeks
  The Fugl-Meyer Assessment scale is to assess the sensorimotor impairment in individuals who have had stroke. The score ranges is 0 to 226. A higher score indicates better body function.
Balance computerized adaptive testing | Baseline to 4 weeks
  The Balance computerized adaptive testing is to assess balance ability.The score ranges is 0 to 10. A higher score indicates better balance ability.
Mini Mental State Examination-2nd edition | Baseline to 4 weeks
  The Mini Mental State Examination-2nd edition is to assess cognitive functions. The score ranges is 0 to 90. A higher score indicates better cognitive functions.
Mini Nutritional Assessment | Baseline to 4 weeks
  The Mini Nutritional Assessment is a comprehensive nutritional assessment scale. The score range is 0 to 30 points. The higher the score, the lower the risk of malnutrition.
Stroke Impact Scale | Baseline to 4 weeks
  The Stroke Impact Scale is to assess health-related quality of life: emotion, communication, memory and thinking, and social role function. The score ranges is 59 to 295. A lower score indicates the quality of life less affected by stroke.
Stroke Self-Efficacy Questionnaire | Baseline to 4 weeks
  The Stroke Self-Efficacy Questionnaire is a self-report scale measuring self-efficacy judgments in specific domains of functioning post stroke. The score ranges is 0 to 130. A higher score indicates better self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: En-Chi Chiu, PhD, Study Director — National Taipei University of Nursing and Health Sciences
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Shihlin District, Taiwan